CLINICAL TRIAL: NCT05825872
Title: Effect of Ultrasound-Guided Internal Superior Laryngeal Nerve Block on Sore Throat After Intubation by Double-Lumen Bronchial Tube for Thoracoscopic Surgery
Brief Title: Ultrasound-Guided Internal Superior Laryngeal Nerve Block for Double-Lumen Bronchial Tube
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, mostafa saieed fahim mansour, lecturer, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2/2023ANET15-1
Record Dates: First submitted 2023-04-11; First posted 2023-04-24 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Postoperative Sore Throat
MeSH Terms: interventions — Lidocaine; Bupivacaine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- control group (No Intervention): patients will undergo a thoracoscopic surgery under general anesthesia with double-lumen bronchial intubation without any special treatment.
- experimental group (Active Comparator): patients will receive US-guided iSLN block bilaterally with 2 ml of ( 0.5 ml of 2%lidocaine and 1,5 ml of 0.5% bupivacaine) on either side immediate after the operation concomitant with GA in order to undergo thoracoscopic surgery
  Interventions: Procedure: internal superior laryngeal nerve block; Drug: Lidocaine 2% Injectable Solution; Drug: Bupivacaine 0.5% Injectable Solution

INTERVENTIONS:
Procedure: internal superior laryngeal nerve block — A linear 4- to 12-MHz ultrasound probe will be placed in the oblique parasagittal plane to obtain an image of the hyoid bone and the thyroid cartilage. The probe will be kept parasagitally, and the following structures will be identified anteriorly to posteriorly: omohyoid muscle, sternohyoid muscle, thyrohyoid muscle, thyrohyoid membrane, superior laryngeal artery, and pre-epiglottis space.
  After identifying the local anatomic structure, a needle will be inserted out-plane from anterior to posterior. The muscles above the thyrohyoid membrane will be penetrated and hydrodissected; local anesthetic will be injected into the superior laryngeal nerve space. The superior laryngeal nerve space will be located between the hyoid bone (cephalad) and the thyroid cartilage (caudal) and delimited between the thyrohyoid muscle, anteriorly, and the thyrohyoid membrane and the pre-epiglottis space, posteriorly
  Arms: experimental group
Drug: Lidocaine 2% Injectable Solution — 0.5 ml will be injected
  Arms: experimental group
Drug: Bupivacaine 0.5% Injectable Solution — 1.5 ml will be injected
  Arms: experimental group

SUMMARY:
investigate the effectiveness and safety of ultrasound-guided bilateral internal branch of the SLN (iSLN) block for alleviating POST immediately after the operation.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1 to 3

Exclusion Criteria:

* patients who did not provide consent
* with a pre-existing sore throat, hoarseness and upper respiratory tract infection
* tracheal pathology, tracheostomy
* a history of psychosis, diabetes and thyroid, oral cavity or pharynx surgery
* known or suspected allergy to ropivacaine
* chronic opioid use
* use of nonsteroidal anti-inflammatory drug medication within 24 hours
* known or suspected difficult airway
* patients who will be supported by tube ventilator after the operation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2023-04-05 (Actual); Primary Completion 2023-07-05 (Estimated); Study Completion 2023-09-05 (Estimated)

PRIMARY OUTCOMES:
the pain classification of postoperative sore throat | from immediate postoperative till 24 hours postoperative
  an established scoring system feom 0 to 4

CONTACTS AND LOCATIONS:
Overall Officials: mostafa s mansour, Study Chair — Menoufia University
Locations (1):
- Menoufia University Hospitals, Shibīn al Kawm, Menoufia, Egypt

IPD SHARING:
Plan to Share IPD: No